CLINICAL TRIAL: NCT05772078
Title: Compliance Rate After Therapy of Peri-implantitis: Retrospective Study
Brief Title: Compliance and Cumulative Interceptive Rate After Therapy of Peri-implantitis
Status: Completed | Type: Observational
Sponsor: Center of Implantology, Oral and Maxillofacial Surgery, Badajoz, Spain (Other)
Responsible Party: Principal Investigator, Alberto Monje, Director, Department of Periodontics, Center of Implantology, Oral and Maxillofacial Surgery, Badajoz, Spain
Other Study IDs: 20230208
Record Dates: First submitted 2023-03-06; First posted 2023-03-16 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2023-10

CONDITIONS: Peri-Implantitis
MeSH Terms: conditions — Peri-Implantitis | interventions — Demography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Compliers: Attending to SPT every 4-6 months
  Interventions: Other: Assess compliance rate and demographics
- Erratic compliers: Attending to SPT once a year or sporadically
  Interventions: Other: Assess compliance rate and demographics
- Non compliers: Non-attenders to SPT
  Interventions: Other: Assess compliance rate and demographics

INTERVENTIONS:
Other: Assess compliance rate and demographics — Records to evaluate attendance rate

SUMMARY:
Peri-implantitis is a plaque-mediated inflammatory condition featured by progressive bone loss. This entity jeopardizes the longevity of dental implants, thus impacting negatively on the quality of life of patients. Moreover, peri-implantitis is suggested to lead to an increased systemic status of inflammation. This may rise the susceptibility to experience life-threating conditions. Therefore, peri-implant infections must be promptly diagnosed and eliminated.

Aiming at resolving the inflammation, several options are advised to remove the infection. Accordingly, implant removal or therapeutic manoeuvres to stablish a healthy ecosystem in the peri-implant environment have been suggested. While the former proved being more predictable, the later demonstrated being more conservative. Indeed, implant removal is commonly associated with regenerative procedures of the alveolar bone deformity that often demand time and is more costly. Anyways, disease severity, implant expendability for biomechanical reasons or esthetic demand seem to be few of the leading aspects in the decision-making process on maintaining or extracting implant showing peri-implant lesions.

Supportive maintenance care (SPT) was shown to be key in preventing disease recurrence. Nonetheless, the compliance of these patients is often erratic. In fact, it is yet unknown the rate of compliance after therapy. Therefore, the goal of this study is to assess the rate and confounders for compliance.

ELIGIBILITY:
Inclusion Criteria:

* Patients that underwent treatment of peri-implantitis
* >12 months of follow-up after therapy
* Patients managed in our center

Exclusion Criteria:

* Patients that were managed in other centers
* Patients that have incomplete records

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients that underwent therapy of peri-implantitis and were recommended to SPT
Sampling Method: Probability Sample
Enrollment: 140 (Actual)
Dates: Start 2023-07-01 (Actual); Primary Completion 2023-07-01 (Actual); Study Completion 2023-10-30 (Actual)

PRIMARY OUTCOMES:
Compliance rate | 1 to 6 years of follow-up
  How many patients are complete compliers

SECONDARY OUTCOMES:
Demographics | 1 to 6 years of follow-up
  Evaluate the patient-related features affecting compliance

OTHER OUTCOMES:
Cumulative Interceptive Rate | 1 to 6 years of follow-upo
  Interventions needed after active therapy to manage peri-implantitis during supportive peri-implant care for erratic and regular compliers

CONTACTS AND LOCATIONS:
Overall Officials: Mamen Tomé, DH, Study Chair — Assistant
Locations (1):
- Centro de Implantologia Cirugia Oral y Maxilofacial, Badajoz, Spain

IPD SHARING:
Plan to Share IPD: Undecided
Publication

REFERENCES:
- [Derived] Monje A, Galindo-Fernandez P, Nart J. Supportive therapy following peri-implantitis treatment: A retrospective study on compliance. Clin Oral Implants Res. 2024 Jun;35(6):621-629. doi: 10.1111/clr.14257. Epub 2024 Mar 26. PMID 38530213